CLINICAL TRIAL: NCT05425134
Title: PET/CT-based Deep Learning Signature for Predicting Occult Nodal Metastasis of Clinical Stage N0 Non-Small Cell Lung Cancer: A Multicenter Prospective Diagnostic Trial
Brief Title: Deep Learning Signature for Predicting Occult Nodal Metastasis of Clinical N0 Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Ningbo No.2 Hospital (Other); Zunyi Medical College (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Chang Chen, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: DLNMS
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer; Lymph node metastasis; Deep learning; PET-CT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/CT-based Deep Learning Signature — Deep Learning Signature Based on PET-CT for Predicting Occult Nodal Metastasis of Clinical N0 Non-small Cell Lung Cancer

SUMMARY:
The purpose of this study is to evaluate the performance of a PET/CT-based deep learning signature for predicting occult nodal metastasis of clinical stage N0 non-small cell lung cancer in a multicenter prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

(1) Participants scheduled for surgery for radiological finding of pulmonary lesions from the preoperative thin-section CT scans; (2) The maximum short-axis diameter of N1 and N2 lymph nodes less than 1 cm on CT scan; (3) The SUVmax of N1 and N2 lymph nodes less than 2.5; (4) Pathological confirmation of primary NSCLC; (5) Age ranging from 20-75 years; (6) Obtained written informed consent.

Exclusion Criteria:

(1) Multiple lung lesions; (2) Poor quality of PET-CT images; (3) Participants with incomplete clinical information; (4) Participants not receiving systematic lymph node dissection; (5) Participants who have received neoadjuvant therapy.

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Clinica N0 Non-small Cell Lung Cancer
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve | 2022.1-2023.12
  Area under the receiver operating characteristic curve

SECONDARY OUTCOMES:
Sensitivity Sensitivity | 2022.1-2023.12
  Sensitivity
Specificity | 2022.1-2023.12
  Specificity
Positive predictive value | 2022.1-2023.12
  Positive predictive value
Negative predictive value | 2022.1-2023.12
  Negative predictive value
Accuracy | 2022.1-2023.12
  Accuracy

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanghai Pulmonary Hospital, Yangpu, Shanghai Municipality
  - Ningbo HwaMei Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No